CLINICAL TRIAL: NCT01146717
Title: Mild Cognitive Impairment:Cerebrovascular Dysfunction and Exercise
Brief Title: Aerobic Exercise Training in Mild Cognitive Impairment Study
Acronym: AETMCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Rong Zhang, Dr. Rong Zhang, UTSW, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 032009-065; R01AG033106-01A2 (NIH)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2016-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; Exercise
MeSH Terms: conditions — Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control group (Placebo Comparator)
  Interventions: Behavioral: Balance training

INTERVENTIONS:
Behavioral: Exercise — Patients with mild cognitive impairment will undergo moderate intensity endurance exercise training for one year.
  Arms: Exercise
Behavioral: Balance training — A group of patients with mild cognitive impairment will perform flexibility and balance training for one year as a control group.
  Arms: Control group

SUMMARY:
This study is being done to find out whether regulation of brain blood flow is altered in patents with mild cognitive impairment (those who have memory problems but otherwise healthy) when compared with healthy elderly individuals. In addition, this study will determine whether exercise training improves brain blood flow, brain structure, and brain function in patients with mild cognitive impairment (MCI).

This is a research study because at present the investigators know little about brain blood flow regulation in patients with mild cognitive impairment. The investigators also know little about whether exercise training improves brain blood flow, brain structure, and brain function in patients with mild cognitive impairment.

DETAILED DESCRIPTION:
We plan to study 70 patients with amnestic MCI and 30 healthy older adults with similar age, sex, and educational level in this research at the University of Texas Southwestern(UTSW) Medical Center Dallas and Texas Health Presbyterian Hospital Dallas - Institute for Exercise an Environmental Medicine (IEEM).

To help decide if you qualify to be in this study, the researchers may ask you questions about your health, including medications you take and any surgical procedures you have had. You may also have to fill out certain forms or have the following exams, tests or procedures. The screening process usually takes 2-3 hours.

You will be required to come for 7-9 visits including the initial screening for eligibility to participate in this study. The experiments will measure your brain perfusion, vascular function and exercise capacity.

For the healthy controls, the expected length of this study will be about 2-3 months including all the test visits. Your participation in this study will end following completion of your testing.

For those with Mild Cognitive Impairment, the expected length of this study will be about 18 months including all the test visits and exercise training. Your participation in this study will end following completion of your repeat testing after one-year exercise training or control intervention. On occasion, training may be delayed due to injury, illness or personal matters. If this is the case, your enrollment in the study may last longer than one year as we attempt to complete the training and testing.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-80 years old, Male or Female
2. Control Subjects: absence of cognitive complaints and normal performance in Uniform Data Set (UDS) neuropsychological tests.
3. For patients: Diagnosis of amnestic MCI (single and multiple domains) by Petersen's criteria (as modified for ADNI-GO study).
4. Stable medical condition for > 6 months
5. Sable medications for >2 months (use of cholinesterase inhibitors, or prior use of multivitamins is allowed)
6. Caregiver/informant available to accompany patient for scheduled visits in case the patient develops cognitive impairment that interferes with independent study participation.
7. Fluency of patient and caregiver in English
8. Ability to return to clinic for additional visits over a 12 month period.
9. ≥ 10 years of education or enough work history to exclude mental retardation.
10. Adequate visual and auditory acuity to allow neuropsychological testing.
11. Screening laboratory tests and ECG without significant abnormalities that might interfere with the study.
12. Physical ability to undergo endurance exercise training.

Exclusion Criteria:

1. Diagnosis of Alzheimer's Disease or other type of dementia.
2. Participant enrolled in any other investigational drug study within 2 months or longer, depending on the investigational drug half-life.
3. Modified Hachinski Score ≥ 4.
4. Subject has history in the past 2 years of epileptic seizures, or DSM-IV criteria of any major psychiatric disorders.
5. Past history or MRI evidence of brain damage including significant trauma, stroke, hydrocephalus, mental retardation or serious neurological disorder.
6. Carotid stent or sever stenosis.
7. Significant history of active alcoholism or drug abuse.
8. History of myocardial infarction within the previous year. Unstable cardiac, renal, lung, liver or other severe chronic diseases.
9. Uncontrolled hypertension (Systolic Blood Pressure (SBP) ≥160, Diastolic Blood Pressure (DBP) ≥100)or hypotension (SBP <100 mmHg).
10. Currently diagnosed and being treated for Diabetes Mellitus (DM).
11. Obesity with Body Mass Index (BMI) ≥ 35.
12. History of familial early onset (<55 years old) dementia
13. Pacemaker or other medical device of metal that precludes performing MRI.
14. Subjects who have been engaged in moderate intensity aerobic exercise training for > 30 minutes, 3 times per week over the past 2 years.
15. History of a clinical diagnosis of B12 deficiency or hypothyroidism. (stable treatment for at least 3 months is allowed).
16. Chronic inflammatory diseases including, lupus, rheumatoid arthritis and polymyalgia rheumatica.

Prohibited Medications:

* narcotics
* anti-Parkinsonian medications
* anti-convulsants for treatment of seizure disorder
* drugs that can influence psychometric test results.

  * Subjects on a statins or non-steroidal anti-inflammatory drug (NSAID) are eligible but must be on a stable dose for at least 2 months.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cognitive function | One year
  A comprehensive battery of neuropsychological tests focused on memory and executive function will be used to assess effects of exercise on cognitive function.

SECONDARY OUTCOMES:
Cerebrovascular function | One year
  Transcranial Doppler and perfusion magnetic resonance imaging (MRI) will be used to measure cerebrovascular function/brain perfusion before and after exercise training.
Brain tissue volume and white matter integrity | One year
  Magnetic resonance imaging (MRI) will be used to measure changes in brain volume and white matter integrity before and after exercise training.

CONTACTS AND LOCATIONS:
Overall Officials: Rong Zhang, PhD, Principal Investigator — UTSW
Locations (1):
- UT Southwestern ADC/Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

REFERENCES:
- [Derived] Pasha EP, Rutjes E, Tomoto T, Tarumi T, Stowe A, Claassen JAHR, Munro Cullum C, Zhu DC, Zhang R. Carotid Stiffness is Associated with Brain Amyloid-beta Burden in Amnestic Mild Cognitive Impairment. J Alzheimers Dis. 2020;74(3):925-935. doi: 10.3233/JAD-191073. PMID 32083583
- [Derived] Stowe AM, Ireland SJ, Ortega SB, Chen D, Huebinger RM, Tarumi T, Harris TS, Cullum CM, Rosenberg R, Monson NL, Zhang R. Adaptive lymphocyte profiles correlate to brain Abeta burden in patients with mild cognitive impairment. J Neuroinflammation. 2017 Jul 27;14(1):149. doi: 10.1186/s12974-017-0910-x. PMID 28750671
- See also: Related Info — http://ieemphd.com/